CLINICAL TRIAL: NCT02259660
Title: Upper Airway Muscle Training for Obstructive Sleep Apnea
Brief Title: Airway Muscle Training for Obstructive Sleep Apnea
Acronym: OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB201400642
Record Dates: First submitted 2014-09-26; First posted 2014-10-08 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; osa; breathing; snoring; respiratory; exercise; inspiratory muscle strength training; expiratory muscle strength training
MeSH Terms: conditions — Sleep Apnea, Obstructive; Respiratory Aspiration; Snoring; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Active Comparator): Subjects in this arm will train their respiratory muscles at home. The training protocol will use progressively higher pressure threshold training valves to provide respiratory muscle strength training at a pressure threshold greater than 70% maximum inspiratory (MIP) and expiratory (MEP) pressures. The total daily training time should be 20 to 30 minutes in duration.
  Interventions: Device: Respiratory muscle strength training
- Sham Training (Placebo Comparator): The intervention in the sham training arm will be identical in every way to that of the active arm with the exception of the trainer that is provided. Subjects in the sham training arm will have inspiratory and expiratory muscle strength trainers which have had the pressure threshold spring removed and are therefore unable to provide a load to the muscles being trained.
  Interventions: Device: Sham respiratory muscle strength training

INTERVENTIONS:
Device: Respiratory muscle strength training — Inspiratory and expiratory muscle strength training occur when subjects are required to breath in (as with inspiratory training) or out (as with expiratory training) through a pressure threshold device. This device features a spring-loaded one way valve which will only open if the subject is able to generate sufficient air pressure to overcome a predetermined pressure threshold. This threshold is typically set at 75% of the subject's maximum capacity. Repeatedly overcoming this threshold during training produces a strengthening effect in most people.
  Other Names: Inspiratory muscle strength training; Expiratory muscle strength training
  Arms: Active Group
Device: Sham respiratory muscle strength training — The placebo / sham intervention will mimic the active intervention(s) in every respect except the devices used will be rendered neutral via removal of the pressure threshold spring inside the devices.
  Other Names: Sham inspiratory muscle strength training; Sham expiratory muscle strength training
  Arms: Sham Training

SUMMARY:
The purpose of this research study is to determine if muscle training will improve snoring and obstructive sleep apnea. Subjects will receive a sleep study to determine the severity of their apnea. After this study, subjects will be randomly assigned to one of two groups. The first group will receiving a breathing trainer that may strengthen the muscles used to breath in and out. The second group will be receive a sham trainer which looks like the "real" trainer but is not able to produce a strengthening effect. Both groups will complete eight weeks of home based (real or sham) training. The sleep study will be repeated and we well measure any changes in measures of severity for obstructive sleep apnea.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disorder characterized by intermittent narrowing or closure of the upper airway during sleep. Loss of muscle tone with sleep onset and decreases in ventilatory drive following the loss of the wakefulness stimuli to breathe combine to result in upper airway closure in patients with structurally susceptible upper airways. We hypothesize that training of upper airway muscles will improve sleep apnea by augmenting the resting upper airway muscle tone and ability of the muscles to respond to negative intraluminal pressure. Training with a primitive wind instrument (such as a Digeridoo) and oral pharyngeal exercises (OPE) used in speech therapy have been shown to improve sleep apnea. Individuals who play certain types of wind instruments appear to have a lower risk of sleep apnea. However, to date the mechanism of improvement and the optimal method of upper airway training have not been well defined. We recently completed a study with a facial exerciser (Facial Flex) designed to improve facial muscle tone and found a decrease in snoring in a group with loud snoring but minimal sleep apnea. A group of UF physiologists (including co investigators Drs. Davenport and Silverman) have also demonstrated that brief periods of training with high inspiratory and/or expiratory threshold loads improved cough and swallowing in patients with impairment in upper airway function. Although respiratory pump muscles provide the driving force for pressure generation during training with pressure threshold loads, the upper airway muscle must maintain a patent upper airway resisting high negative or positive intraluminal pressures. For example, the palate must maintain a seal preventing air escape through the nose when high positive pressure is generated through a mouthpiece. Of interest a limited number of very high intensity efforts appears to be the optimal way to train muscles.

We propose targeting a group of mild to moderate OSA patients (apnea-hypopnea index < 30/hour) who are not severely obese (BMI < 35 Kg/M2) and do not have significant structural abnormalities of the upper airway or muscle dysfunction. We will perform a randomized controlled trial (training versus sham training) with 25 subjects in each treatment arm using two months of daily training (5 out of 7 days each week). A home sleep study (including EEG) will be performed before and following the training. The change in the apnea-hypopnea index adjusted for sleep stage and body position will be compared. Use of home sleep studies will dramatically reduce the cost of the study. A sleep technologist will educate subjects on performance of maneuvers and meet with them weekly to observe the subject's technique. A training log will be kept by the subjects using training schedule sheets and daily training will be monitored through weekly web-based communication with a study clinician.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* AHI ≥ 5/hour and less than 30/hour
* Ability to understand and perform training.
* Ability to return to the UFHealth Sleep Center 1X per week for the (8 week) duration of the study.

Exclusion Criteria:

* Pregnancy
* Prior Upper airway surgery (nasal surgery is allowed)
* Severe nasal obstruction
* BMI > 35 kg/M2
* Use of potent narcotics
* History of arrhythmia (other than PACs and PVCs)
* Coronary artery disease or congestive heart failure (patients with controlled hypertension will be included),
* Moderate to severe lung disease
* History of pneumothorax.10. severe daytime sleepiness (falling asleep while driving or
* Epworth Sleepiness Scale [Appendix 1] > 14),
* History of chronic short sleep duration (< 5 hours).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09-28 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | Baseline and 10 weeks
  The AHI is a measure of symptom severity for obstructive sleep apnea. Physiological data obtained during a sleep study is used to complete this measure.

SECONDARY OUTCOMES:
Maximum inspiratory pressure (MIP) | Baseline and 10 weeks
  MIP is an estimate of the strength of respiratory muscles that are used to inhale. Specifically, the diaphragm and external intercostals. This measure is obtained by having the subject inhale forcibly through a mouthpiece connected to a pressure manometer.
Maximum expiratory pressure (MEP) | Baseline and 10 weeks
  MEP is an estimate of the strength of breathing muscles used for exhalation. Specifically, the abdominals and internal intercostals. MEP is obtained by having the subject exhale forcibly through a mouthpiece that is connected to a pressure manometer.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Berry, M.D., Principal Investigator — University of Florida
Locations (1):
- UFHealth Sleep Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided